CLINICAL TRIAL: NCT07079787
Title: Telerehabilitation of Balance Clinical and Economic Decision Support System
Brief Title: Telerehabilitation Decision Support System: Pilot Testing Protocol
Acronym: TeleRehab DSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University Medical Center Freiburg (Other); King Chulalongkorn Memorial Hospital (Other); Secretaria Regional de Saúde e Proteção Civil da Região Autónoma da Madeira (Unknown); Institute of Communications and Computer Systems, Athens, Greece (Other); University of Ioannina (Other); Vilabs (Unknown); BioIRC (Unknown); Activage (Unknown); Institue De Desenvolvimento De Novas Technologiassociacao (Unknown); Quantitas SRL (Unknown); Instituto para o Desenvolvimento e Inovação (Unknown); BRIDG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCLondon17413/002
Record Dates: First submitted 2025-06-30; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Mild Cognitive Impairment (MCI); Vestibular Disease; Long Covid-19
Keywords: vestibular; rehabilitation; falls; balance; exercise; artificial intelligence; teleremedicine; physiotherapy
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Vestibular Diseases; Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: In this pilot testing study, participants will be blinded to their allocation gorup, but due to the nature of the study, assessors will not be. Participants will be randomised by condition (stroke, MCI, long covid-19, vestibular disorders) into either the high-technolog or low-technology solution and will carry out the intervention under the supervision of the assessing clinician.
Who Masked: Participant
Masking Description: Participants will be blinded to which study arm participants have been allocated to. Due to the nature of the study, the assessing and treating clinician cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Technology (Active Comparator): All TeleRehab DSS components: multisensory balance exercises, AR avatar, real-time feedback, AR gamified activities, sensor-monitored exercise performance, and additional cognitive training.
  Interventions: Device: TeleRehab DSS Pilot Test
- Low-Technology (Active Comparator): With depth camera, motion sensors and tablet for multisensory balance exercises, real time feedback, sensor monitored exercise performance and cognitive games. No exergames, no smartwatch, no mobile phone.
  Interventions: Device: TeleRehab DSS Pilot Test

INTERVENTIONS:
Device: TeleRehab DSS Pilot Test — Participants will perform an individualised multisensory balance rehabilitation program via augmented reality, while wearing motion sensors. The program will consist of multisensory balance exercises, cognitive games, and exergames. All participants will perform 2 sessions per week, carried in at each clinical site, over the course of 3-week.s

SUMMARY:
This study follows the successfully completed HOLOBalance project which was funded by the EU Horizon 2020 scheme. TheHOLOBalance platform delivers exercises demonstrated via a hologram of the physiotherapist and corrected in real time by the hologram prompts based on performance monitoring via sensors. Further information is available at: https://holobalance.eu/. HOLOBalance was developed as a comprehensive rehabilitation protocol for individualised remote (tele)rehabilitation balance physiotherapy programme. It includes different multisensory balance and gait exercises, physical activity and memory training and exergames (video games which are also exercises) to improve balance function in older adults. The system can thus assess and remotely monitor how users are performing the exercises.

This pilot testing of a multisite randomised control trial (TeleRehab DSS, short for TeleRehabilitation Decision Support System) aims to investigating the usability and feasibility among a smaller sample population at each clinical site, identifying any technical bugs, and/or clinical procedural flaws to be remedied before delivery of the full-scale RCT.

DETAILED DESCRIPTION:
This is a multi-centre pilot study to test the usability and feasibility of the TeleRehab DSS platform among a sample population across all five clinical sites.

Upon meeting the initial inclusion criteria, eligible participants will be scheduled for an appointment to attend the clinic and complete a cognitive assessment (MoCA) and gait assessment (FGA). If a participant is deemed fully eligible, they will proceed with the onboarding process and clinical assessment, including the collection of personal details and a set of health questionnaires. They will then be randomised into either the high-tech or low-tech TeleRehab DSS intervention group.

All study participants will attend two sessions weekly over 3-weeks at each clinical site, where they will complete a personalised multisensory balance rehabilitation programme using augmented reality while wearing motion tracking sensors. Clinicians will be present to attend to any technical or clinical queries during completion of the program. At the end of the 3-weeks, the artifical intelligence decision support system will suggest exercise progressions, tracking wether the clinical agrees or disagrees with these suggestions.

Participants will receive telephone calls each week to monitor their progress. Participants will also receive remote program reviews at weeks 3, 6 and 9, from a member of the research team to assess and change exercises as required. Participants will be advised to contact the research team by email or by telephone during working hours if they have concerns or questions about their rehabilitation program or the TeleRehab DSS system. The research team will judge whether an additional home visit is required. If a patient does not complete their exercises for three consecutive days, a flag/warning will appear on the patients dashboard as a priority patient to follow up with, within 24 hours.

TeleRehaB DSS supported, prescribed, progressed and delivered intervention. In the TeleRehaB DSS IG, the platform will suggest two possible management strategies, on an individualised basis, based on patient profiles and expected benefit: 1)The high-tech, full TeleRehaB DSS with all components of the intervention consisting of TeleRehaB DSS AI-progressed multisensory balance exercises with the use of the AR avatar, real time feedback, AR gamified intervention, sensor monitored exercise performance and additional cognitive training, 2) the low-tech, basic version of TeleRehaB DSS, with depth camera, sensors and tablet - multisensory balance exercises, real time feedback, sensor monitored exercise performance and cognitive games, with no exergames, no smartwatch, and no mobile phone. The clinician can override the TeleRehab DSS group allocation decision if it is deemed unsafe.

ELIGIBILITY:
ALL PARTICIPANT Inclusion Criteria:

* Age 40-80 years
* community dwelling able to walk 500-m independently or with a stick
* Depression subscale on Hospital Anxiety and Depression Scale <10/21 (14-item questionnaire)
* No significant visual impairment (as self-reported by participants)
* Willing to comply with study procedures, proposed training and testing regime
* With capacity to consent
* No acute musculoskeletal or other injuries that would prevent participation in a structured exercise program
* Is not currently, and has not in the past 8-weeks received any falls/balance/vestibular and/or cognitive rehabilitation.
* Does not any implanted medical devices or a cardiac pacemaker.
* Does not have any other co-existing neurological conditions (ie. Multiple sclerosis, Parkinson's disease, neuropathy etc.)
* Does not have any language or communication deficits impairing their ability to communicate and/or express their thoughts.
* Has at least one functional hand for grip function and computer use.
* Fulfilling all of the criteria from one of the below sub-groups

STROKE COHORT who will fulfil the additional criteria:

* Individuals with diagnosis of focal ischaemic or haemorrhagic stroke, as confirmed by a clinical letter.
* Onset >/= 3 months prior to study.
* Montreal Cognitive Assessment (MoCA) score n >/=23
* At risk of falls (i.e. Functional Gait Assessment FGA score </=22/30; FGA is a validated quick balance task assessment) AND/OR having experienced a fall(s) in the last 12 months

MCI COHORT who will fulfil the additional criteria:

* Individuals with new or existing formal diagnosis of MCI, according to the International Classification of Disease 10 (ICD10) , as confirmed by a clinical letter.
* At risk of falls (FGA </= 22/30) AND/OR having experienced a fall(s) in the last 12 months.

VESTIBULAR COHORT who will fulfill the additional criteria

* Montreal Cognitive Assessment (MoCA) score n >/=23
* Individuals with a diagnosis of a vestibular disorder (peripheral and/or mixed peripheral and central):
* Peripheral vestibular disorder in which the balance problem lies in the vestibular/balance system within the inner ear.
* Mixed vestibular disorder in which the balance problem lies in the vestibular/balance system within the inner ear (peripheral) and involving the nerves or neuronal network in the brain/brainstem responsible for balance (central).
* Chronic dizziness and/or unsteadiness (>/= 3 months duration) that started at the time or after the vestibular disorder diagnosis.
* Dizziness handicap inventory (DHI >34) AND/OR At risk of falls (FGA </=22/30)

LONG COVID-19 COHORT who will fulfill the additional criteria:

* Montreal Cognitive Assessment (MoCA) score n >/=23
* Individuals with laboratory confirmed diagnosis of Covid (>/=6 months prior to study onset), as confirmed by a clinical letter.
* Who have been diagnosed with long Covid, as confirmed by a clinical letter.
* Who have chronic dizziness and/or unsteadiness which started after the Covid illness (self-report by the patient; duration </=3 months).
* Dizziness handicap inventory (DHI >34) AND/OR At risk of falls (FGA </=22/30)

Exclusion Criteria:

* Outside of the stated age bracket
* Unable to walk independently (even with use of a walking stick)
* MOCA score <23
* Score of 10 or higher on depression subscale of HADS
* Unwilling to comply with study procedures, proposed training and testing regime
* No capacity to consent
* Significant visual impairment or homonymous hemianopia (stroke cohort only) (self-reported)
* Orthostatic hypotension or uncontrolled hypertension
* Other neurological problem (e.g. Parkingson's disease, Multiple Sclerosis etc.)
* Language and communication deficits impairing ability to express thoughts (e.g. Aphasia)
* Has participated in a clinical drug trial in the past 6 months.
* Acute musculoskeletal injury that prevents participation in a structured exercise programme (e.g. lower limb fracture).
* Has an implanted medical device or cardiac pacemaker.
* Diagnosis of unstable Meniere's or with more than 4 migraines/month at the time of participating in the study
* Not fulfilling the inclusion criteria for one of the sub-groups (such as criteria for Stroke group, or MCI group, or chronic vestibular disorder group, or long-Covid group), as outlined above.
* Unable to provide a clinical letter confirming diagnosis.
* For those with stroke, no visual spatial neglect.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety) | Baseline assessment (week 1) through to the last session of Week 3
  Participants will be monitored for adverse events during telephone or face-to-face contacts as part of the intervention phase and during follow-up assessments. Any adverse events related to the treatment will be reported via an adverse events form on the system database. Falls diaries will be collected weekly from participants during the intervention and monthly for up to 6 months after completion of the intervention.
Recruitment Rate (acceptability) | Baseline assessment (week 1) through to the last session of Week 3
  percentage of recruited participants that were eligible
Feasibility (protocol deviations/problems) | Baseline assessment (week 1) through to the last session of week 3
  Incidence of protocol deviation and/or implementation problems reported during the intervention.
Participants experience using the system (usability) | Baseline assessment (week 1) through to the last session of week 3
  Participants experience using the system gathered via qualitative feedback throughout the testing period and post-intervention via exit interviews
Adherence to Intervention | Week 1 through to completion at week 3
  percentage of prescribed sessions completed throughout the intervention
Drop-out rate (acceptability) | Baseline (week 1) through to last session in week 3
  Percentage of enrolled participants that were loss to follow-up or drop-outs

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | Baseline assessment through to the last session of Week 3
  test that assesses complex gait tasks (e.g. walking with head turns or stopping and turning, 5 minutes).
Mini Balance Evaluation Systems Test (Mini-BESTest) | Baseline assessment through to the last session of Week 3
  a 14-item test that assesses dynamic balance, on a scale of 0 (indicating severe balance impairment) to 28 (representing normal balance with a total score of 28 points).
Montreal Cognitive Assessment (MoCA) | Baseline assessment through to the last session of Week 3
  includes sections on visuospatial/executive function, naming, attention, language, abstraction, memory and orientation to time and place (6 questions) with a scor range from 0-30, with a higher score indicating better cognitive function.
EuroQol five dimensional descriptive system (EQ-5D-5L) | Baseline assessment through to the last session of Week 3
  Measure of quality-adjusted life years (QALYs). EQ-5D-5L is a standardized, valid and reliable simple, generic measure of health status for clinical and economic appraisal. The respondent is asked to rate their health status on these five dimensions from 1 to 5 respectively as no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS (Visual Analogue Scale) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The respondent is asked to mark an X on the scale to indicate "how your health is TODAY" with a higher score indicating better health-related quality of life
Rapid Assessment of Physical Activity (RAPA) | Baseline assessment through to the last session of Week 3
  The 9-item self-administered Rapid Assessment of Physical Activity (RAPA) is a questionnaire that assesses levels of a wide range of physical activity level in adults older than 50 years, with a score range 1-7 and a higher score indicating ihgher levels of physical activity.
Dizziness Handicap Inventory (DHI) | Baseline assessment through to the last session of Week 3
  The 25-item self-report Dizziness Handicap inventory (DHI) validated questionnaire that assesses functional, emotional and physical domains. Responses are graded 0 (no), 2 (sometimes) or 4 (yes) with higher scores indicating greater impact of dizziness maximum and maximum score of 100 points (15 minutes).
The Activities-specific balance confidence scale (ABC) | Baseline assessment through to the last session of Week 3
  The Activities-specific Balance Confidence Scale (ABC) that assesses patient's perceived confidence for 16-activities of daily living without losing balance .Score range from 0-100 with higher schore indicating greater balance confidence and scores ≤67/100% indicate increased falls risk.
The Hospital Anxiety and Depression Scale (HADS-d) depression subscale | Baseline assessment through to the last session of Week 3
  14-item scale which assesses non-somatic anxiety (HAD-A) and depression (HAD-D) symptoms. Scores range from 0-21 for each subscale, with higher scores indicating worse outcomes (greater anxiety or depression).
Fatigue Severity Scale (FFS) | Baseline assessment through to the last session of Week 3
  a 9-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them. Sca;e 9-63 with higher score indicating greater fatigue.
Warwick-Edingburgh Mental Wellbeing Scale (WEMWBS) | Baseline assessment through to the last session of Week 3
  developed to enable the measuring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing. The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing, thereby making the concept more accessible. The scale has been widely used nationally and internationally for monitoring, evaluating projects and programmes and investigating the determinants of mental wellbeing. Scale 14-70 with higher score indicating better mental wellbeing.
Situational Vertigo Questionnaire (SVQ) | Baseline assessment through to the last session of Week 3
  The SVQ is 20-item questionnaire designed to assess discomfort in situations of intense visual salience of visual-vestibular conflict. It was originally developed as a measure of space and motion discomfort. The questions are graded on a scale from 0 (not at all) to 4 (very much), with a higher score indicating greater vertigo severity.
The system Usability Scale (SUS) | Post-intervention (end of Week 3)
  The System Usability Scale (SUS) scale 1-5 rated on 10 aspects, with a total possible score of 0-100, with a higher score indicated better usability.
User experience questionnaire (UEQ) | Post-intervention (end of Week 3)
  he User Experience Questionnaire (UEQ; scale 1-7 on 26 dimensions of attractiveness, perspicuity, efficiency, dependability, stimulation and novelty with a score range of -3 (worst) to +3 (best) with a higher score indicating a more positive user experience.

OTHER OUTCOMES:
Falls | collected weekly for the duration of the 3-week intervention
  Occurence of falls, and reasoning if any falls took place, self-reported via a falls diary.
System performance | post-intervention (week 3)
  We will also compare the TeleRehaB DSS predicted versus observed patient outcomes on the EQ-5D-5L, and secondary outcome measures, to assess the system performance
eHealth Literacy Assessment (eHEALS) | Baseline (week 1)
  a 10-item likert scale questionnaire that evaluate's patients' skills in finding, evaluating and applying electronic health information. Responses range from 1 (strongly disagree, to 65 (strong agree), with total scores indicating levels of eHealth literacy. This will be used to help validate the AI-model in terms of participant allocation into the high-tech versus low-tech solution.
The Senior technology acceptance & adoption model (STAM) | Baseline (week 1)
  is a 38-item questionnaire, with items rated on a 1-10 Likert scale to measure factors influencing technology acceptance among older adults, with a higher scores indicating greater perceived digital literacy.
Mobile Device Proficiency Questionnaire - short (MDPQ-s) | Baseline (week 1)
  is a 16-question version of the full MDPQ-16. The MDPQ, its subscales, and the MDPQ-16 were found to be highly reliable and valid measures of mobile device proficiency in a large sample. We conclude that the MDPQ and MDPQ-16 may serve as useful tools for facilitating mobile device training of older adults and measuring mobile device proficiency for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, PhD, Principal Investigator — University College, London
Locations (5):
- University Medical Center Freiberg Neurocenter (UKLFR), Freiberg,, Freiburg im Breisgau, Germany
- National and Kapodistrian University of Athens, Athens, Greece
- Secretaria Regional de Saúde e Proteção Civil da Região Autónoma da Madeira, Madeirã, Portugal
- King Chulalongeorn Memorial Hospital, Bangkok, Thailand
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data collected will be analysed for improving the system ahead of the full-scale RCT. No participant identifiable data will be included in the final study reports or in the process of dissemination of the study results. The participants will be guided to where they can access the final result publication(s). Anonymised data will be stored securely in an encrypted dashboard and data repository and will be available to other project members and other researchers in line with open science. The research data collected in the course of the study will be retained by UCL and other clinical partners in their capacity as a sponsor for 20 years after the research study has ended. The data will be then securely destroyed.
Supporting Information: Study Protocol, ICF
Time Frame: 20 years after the research study has ended; July 2026 - July 2046
Access Criteria: All study research team members at all clinical sites will comply with their local requirements with regards to the collection, storage, processing and disclosure of personal information and will uphold the Act's core principles.
  The creation of coded, depersonalised data where the participant's identifying information will be replaced by an unrelated sequence of characters will be in place. The digital data collected will be stored in digital format at each clinical sites secure safe haven data platform with encrypted and password protection. The data (hard copies) collected during the study will be stored in the study site file in a securely locked designated cabinet at each clinical site for the duration of the study.